CLINICAL TRIAL: NCT05156229
Title: A Phase 1/2a Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneously Administered CDK-003 in Healthy Adult Participants and Intralesionally Administered CDK-003 in Patients With Cutaneous T-cell Lymphoma (CTCL)
Brief Title: A Phase 1/2a Study of CDK-003 in Patients With Cutaneous T-Cell Lymphoma (CTCL).
Acronym: Part B
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PK/PD from two patients plus the healthy volunteer data confirmed the RP2D and manageable safety profile. Proceeding to Phase II did not require additional data from this Phase I Dose-Finding study.
Sponsor: Codiak BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDK-003-101
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Cutaneous T-cell Lymphoma (CTCL)
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CDK-003 (Experimental): CDK-003 administered subcutaneously every 2 weeks.
  Interventions: Biological: CDK-003

INTERVENTIONS:
Biological: CDK-003 — CDK-003 administered subcutaneously

SUMMARY:
This is a Phase 1, dose escalation study to assess the safety, tolerability, pharmacokinetic and pharmacodynamic effects of CDK-003. The study is performed in two parts: Part A is a randomized, double-blind, placebo-controlled, single ascending dose study of CDK-003 in healthy adult male participants, and Part B is a single arm, open-label, multiple ascending dose in patient-participants with CTCL. Dose escalation in the study will only occur after satisfactory review of all available predefined data by the Safety Review Committee. Part A is complete and this entry describes Part B only.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed CTCL as per Olsen et al, 2011 or per algorithm for diagnosis of early MF as per Pimpinelli et al, 2005.
2. Patient-participants with Stage IA-IIB CTCL (MF) with injectable lesions (patches, plaques, or tumors), who have relapsed or refractory disease following at least 1 prior standard treatment. Patient-participants who are unsuitable to receive standard treatment or who have declined standard treatment are also eligible.
3. Patient-participants must have ≥ 1 treatable/measurable lesion(s) for injection as per Olsen criteria.
4. Understands and is able to comply with the study requirements and has signed the informed consent form.
5. Has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
6. Life expectancy of at least 6 months.
7. Age 18 years or older at the time of signing the informed consent form.
8. Acceptable liver function:

   1. Bilirubin equal 1.5x ULN.
   2. AST (SGOT), ALT (SGPT) equal 3.0x ULN.
9. Acceptable renal function:

   a. Serum creatinine ≤ 1.5x ULN.
10. Acceptable hematologic status:

    1. Absolute neutrophil count - 1500 cells/mm3
    2. Platelet count - 100,000 /mm3
    3. Hemoglobin - 9 g/dL.
11. Acceptable coagulation status: international normalized ratio ≤ 1.5 ULN. Patient-participants on therapeutic doses of vitamin K antagonists (eg, warfarin) or direct oral anticoagulants (eg, direct thrombin or direct factor Xa inhibitors) are not eligible.

    Anticoagulation with low molecular weight heparins is permitted.
12. Women of child-producing potential agree to use highly effective contraceptive methods (see Appendix C for details) for one complete menstrual cycle (or at least 30 days) prior to the first dose of CDK-003 until 6 months following the last dose of CDK-003, and avoid egg donation from the time of the first dose of CDK-003 until 6 months following the last dose of CDK-003. A female participant is considered to be of child-producing potential unless she:

    1. has had a hysterectomy or bilateral oophorectomy or
    2. is age ≥ 60 years and is amenorrhoeic or
    3. is age < 60 years and has been amenorrhoeic for ≥ 12 months (including no irregular menses or spotting) in the absence of any medication which induces a menopausal state and has documented ovarian failure by serum estradiol and follicle-stimulating hormone levels within the institutional laboratory postmenopausal range).
13. A negative pregnancy test (if a woman of child-producing potential) within 72 hours prior to the first dose of CDK-003.
14. Men of child-producing potential agree to use highly effective contraceptive methods and avoid sperm donation from the time of the first dose of CDK-003 until 6 months following the last dose. Male patient-participants must use a condom when engaged in intercourse during the study and for 6 months after the last dose of study drug.

    A man is considered to be of child-producing potential unless he has had a bilateral vasectomy with documented aspermia or a bilateral orchiectomy.
15. Patient-participant agrees to have a pre-treatment tumor biopsy during the Screening Period, and 2 on-treatment tumor biopsies of the same lesion.

Exclusion Criteria:

1. Patient-participants with CTCL disease involving N3 nodes.
2. Clinically significant ongoing AEs that have not returned to baseline or to Grade 1 National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 during the Screening Period.
3. Received nitrogen mustard, PUVA, narrow band UVB light therapy, carmustine (BCNU), other systemic therapies, radiation therapy or investigational agents for CTCL within 21 days of Day 1.
4. Received systemic corticosteroids within 28 days of Day 1.
5. Use of topical corticosteroids on any of the target lesions for CDK-003 injection or non-injected target lesion within 28 days of Day 1. Topical corticosteroid use is permitted for non-target lesions.
6. Major surgery within 2 months or minor surgery (excluding tumor biopsies) within 14 day prior to Day 1.
7. Clinically significant cardiovascular disease including but not limited to myocardial infarction or stroke within the past 6 months prior to Day 1, New York Heart Association Class III or IV heart failure, uncontrolled arrhythmia, or severe aortic stenosis. Sponsor approval of patient-participants with an arrhythmia is required.
8. Active, uncontrolled bacterial, viral, or fungal infections requiring systemic therapy.

   Prophylactic antibiotics are acceptable.
9. Prior organ or stem cell transplant.
10. Primary immune deficiency.
11. Pregnant or nursing women.
12. Positive test for HBsAg, HCV Ab, or HIV Ab during the Screening Period.
13. Unwillingness or inability to comply with procedures required in this protocol.
14. Serious non-malignant disease (e.g., liver failure, ongoing infection requiring intravenous treatment, psychological illness, autoimmune disease including but not limited to inflammatory bowel disease, or other conditions) or social situations that, in the opinion of the Investigator and/or the Sponsor, could compromise protocol objectives or patient participant safety or the ability of the patient-participant to comply with the protocol.
15. History of another malignancy, unless potentially curative treatment has been performed. Sponsor approval is required. Patient-participants with early stage prostate cancer on active surveillance may be enrolled with Sponsor approval.
16. Currently receiving any other anti-cancer or investigational agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | up to 2 years
  To determine the safety, tolerability, and DLTs of CDK-003 monotherapy following multiple ascending dose escalation in patient-participants with CTCL
Primary Outcome | up to 2 years
  To identify a recommended phase 2 dose (RP2D) for CDK-003 monotherapy.

SECONDARY OUTCOMES:
Secondary Outcome | up to 2 years
  To evaluate the preliminary anti-tumor activity of CDK-003 monotherapy

OTHER OUTCOMES:
Exploratory Outcome | up to 2 years
  To evaluate potential pharmacodynamic biomarkers associated with treatment with CDK-003 monotherapy that may correlate with any anti-tumour effect.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Scarisbrick, MD, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - University Hospital Birmingham, Birmingham
  - Beatson West of Scotland Cancer Centre Haematology, Glasgow
  - Guys Hospital/ Guy's Cancer Centre, London
  - The Christie, Manchester

IPD SHARING:
Plan to Share IPD: No